CLINICAL TRIAL: NCT02829957
Title: Randomized Trial to Test the Effect of Rivaroxaban or Apixaban on Menstrual Blood Loss in Women
Brief Title: RAMBLE - Rivaroxaban vs. Apixaban for Heavy Menstrual Bleeding
Acronym: (RAMBLE)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jeffrey Kline, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMBLE; NCT02761044 (obsolete NCT alias)
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Venous Thromboembolism; Menstruation
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Active Comparator)
  Interventions: Drug: Rivaroxaban
- Apixaban (Active Comparator)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — 10mg BID for 7 days, then 5mg BID for three months
  Other Names: Eliquis
  Arms: Apixaban
Drug: Rivaroxaban — 15mg BID for 7 days, then 20mg daily for three months
  Other Names: Xarelto
  Arms: Rivaroxaban

SUMMARY:
A large proportion of women with menstruating potential with newly diagnosed VTE or atrial fibrillation, treated with apixaban will have less menstrual blood loss than patients randomized to rivaroxaban.

DETAILED DESCRIPTION:
Heavy menstrual bleeding (HMB) complicates the treatment of approximately 9-25% of patients treated with orally administered anti-Xa anticoagulants for venous thromboembolism (VTE, including either pulmonary embolism or deep vein thrombosis). In particular, recent evidence has suggested an increase in length and severity of menstrual bleeding for women treated with rivaroxaban, and this effect may be less severe apixaban treatment.(1;2) Increase in uterine bleeding with rivaroxaban has necessitated hysterectomy in rare cases.(3) Other complications of HMB include reduced drug adherence, decreased perception of wellness (quality of life) and anemia.(4;5) The anti-Xa agents may increase HMB more than vitamin K antagonists.(1) However, in the principal investigators' experience treating over 100 women of menstruating age with rivaroxaban for VTE with varying degree of HMB, no woman has expressed desire to switch to a VKA even when offered this option (unpublished data). We have successfully reduced perception of HMB by switching from rivaroxaban to apixaban in six patients. Comparison of published and supplemental data from AMPLIFY and AMPLIFY Extend to EINSTEIN and EINSTEIN extend trials also support a lower rate of uterine bleeding with apixaban compared with rivaroxaban, although exact comparisons are difficult to make.(6;9) Myers et al recently reported a 9.4% rate of HMB with apixaban, compared with a 25% rate of HMB with rivaroxaban.(2) Accordingly, we hypothesize that women with menstruating potential with newly diagnosed VTE or atrial fibrillation/flutter, treated with apixaban will have less menstrual blood loss than patients randomized to rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women, age 18-50

  * For study purposes, evidence of negative pregnancy is accounted for by the treating physician's initiation of treatment with oral anticoagulants
* Objectively diagnosed VTE or atrial fibrillation/flutter
* Patient reported active menstruation - does not apply to women who were recently pregnant
* Clinical plan and patient agreement to treat with oral anticoagulation for 3 months or longer
* Patients must have a working telephone

Exclusion Criteria:

* Package insert exclusions for Eliquis (Apixban) or Xarelto (Rivaroxaban): [active pathological bleeding or severe hypersensitivity reaction to XARELTO or ELIQUIS (e.g., anaphylactic reactions)]
* Plan to become pregnant in the next three months.
* Concomitant prescribed use of aspirin or thienopyridenes or other platelet inhibiting drugs
* Plan for surgical hysterectomy or endometrial ablation
* Known uterine cancer
* Von Willebrand's disease, or hemophilia
* Known coagulopathy from liver disease
* Conditions likely to preclude adherence to study procedures: Active intravenous drug use, known alcoholism, homelessness, or uncontrolled psychiatric illness.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09; Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Kline, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Health System, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana

REFERENCES:
- [Background] De Crem N, Peerlinck K, Vanassche T, Vanheule K, Debaveye B, Middeldorp S, Verhamme P, Peetermans M. Abnormal uterine bleeding in VTE patients treated with rivaroxaban compared to vitamin K antagonists. Thromb Res. 2015 Oct;136(4):749-53. doi: 10.1016/j.thromres.2015.07.030. Epub 2015 Aug 4. PMID 26272306
- [Background] Myers B, Webster A. Heavy menstrual bleeding on Rivaroxaban - Comparison with Apixaban. Br J Haematol. 2017 Mar;176(5):833-835. doi: 10.1111/bjh.14003. Epub 2016 Mar 11. No abstract available. PMID 26970315
- [Background] Beam DM, Kahler ZP, Kline JA. Immediate Discharge and Home Treatment With Rivaroxaban of Low-risk Venous Thromboembolism Diagnosed in Two U.S. Emergency Departments: A One-year Preplanned Analysis. Acad Emerg Med. 2015 Jul;22(7):788-95. doi: 10.1111/acem.12711. Epub 2015 Jun 25. PMID 26113241
- [Background] Kline JA, Kahler ZP, Beam DM. Outpatient treatment of low-risk venous thromboembolism with monotherapy oral anticoagulation: patient quality of life outcomes and clinician acceptance. Patient Prefer Adherence. 2016 Apr 15;10:561-9. doi: 10.2147/PPA.S104446. eCollection 2016. PMID 27143861
- [Background] Liu Z, Doan QV, Blumenthal P, Dubois RW. A systematic review evaluating health-related quality of life, work impairment, and health-care costs and utilization in abnormal uterine bleeding. Value Health. 2007 May-Jun;10(3):183-94. doi: 10.1111/j.1524-4733.2007.00168.x. PMID 17532811
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- [Background] EINSTEIN Investigators; Bauersachs R, Berkowitz SD, Brenner B, Buller HR, Decousus H, Gallus AS, Lensing AW, Misselwitz F, Prins MH, Raskob GE, Segers A, Verhamme P, Wells P, Agnelli G, Bounameaux H, Cohen A, Davidson BL, Piovella F, Schellong S. Oral rivaroxaban for symptomatic venous thromboembolism. N Engl J Med. 2010 Dec 23;363(26):2499-510. doi: 10.1056/NEJMoa1007903. Epub 2010 Dec 3. PMID 21128814
- [Background] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivaroxaban | Apixaban
Started | 8 | 11
Completed | 6 | 10
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: The number of participants at baseline differ from those of the outcome measurements because some participants were lost to followup.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Apixaban | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19
d-dimer [Median (Full Range); unit: ng/ml] — D-Dimer normal level < 250
  ng/ml | 661 [327 to 1176] | 1031 [404 to 49815] | 840.5 [327 to 49815]
pbac-pictoral bloodloss assessment chart [Median (Full Range); unit: score] — A PBAC Score of < 100 indicates a normal menstrual cycle. The lowest possible score would be zero. Higher values indicate worse outcomes. The higher theoretical range value cannot be calculated. The scoring mechanism is as follows;
  Towels
  1 point for each lightly stained towel 5 points or each moderately soiled towel 20 points if the towel is completely saturated with blood
  Tampons 1 point for each lightly stained tampon 5 points for each moderately soiled tampon 10 points if the tampon is completely saturated with blood
  Clots
  1 point for small clots 5 points for large clots
  score | 173.5 [39 to 785] | 142 [74 to 320] | 148 [39 to 785]
hgb [Median (Full Range); unit: g/dl] — Normal hemoglobin range for adult women - 12 - 16 g/dL. Lower levels indicate worse outcomes.
  g/dl | 12.6 [11.4 to 14.7] | 13.0 [7.1 to 15.0] | 12.7 [7.1 to 15.0]
Short Form Health Survey (SF-36) [Median (Full Range); unit: Score] — The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
  Score | 57.9 [35.4 to 75.4] | 55.4 [25.8 to 80.6] | 55.4 [25.8 to 80.6]

OUTCOME MEASURES:

1. Primary Outcome: PBAC Scores
Description: Measure Description: A PBAC Score of < 100 indicates a normal menstrual cycle. The lowest possible score would be zero. Higher values indicate worse outcomes. The higher theoretical range value cannot be calculated. The scoring mechanism is as follows;
  Towels
  * 1 point for each lightly stained towel
  * 5 points or each moderately soiled towel
  * 20 points if the towel is completely saturated with blood
  Tampons
  * 1 point for each lightly stained tampon
  * 5 points for each moderately soiled tampon
  * 10 points if the tampon is completely saturated with blood
  Clots
  * 1 point for small clots
  * 5 points for large clots
Time Frame: 3 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 6 | 10
score on a scale | 292 [74 to 600] | 146 [3 to 378]

2. Secondary Outcome: Number of Participants Who Discontinued Planned Drug Administration
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 8 | 11
Participants | 4 | 2

3. Secondary Outcome: Number of Patients That Held Drug for Menorrhagia
Time Frame: 1, 2, and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Major Hemorrhage
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Venous Thromboembolism (VTE)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 8 | 11
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Who Crossed Over to Another Anticoagulant
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 8 | 11
Participants | 3 | 1

7. Secondary Outcome: Number of Participants With Clinically Relevant Non-major Bleeding
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 8 | 11
Participants | 3 | 0

8. Secondary Outcome: Hemoglobin Concentration
Description: Measure Description: Normal hemoglobin range for adult women - 12 - 16 g/dL. Lower levels indicate worse outcomes.
Time Frame: 3 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: g/dl
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 4 | 10
g/dl | 12.8 [11.6 to 14.5] | 13.25 [10.7 to 14.6]

9. Secondary Outcome: Physical Component Summary of Standard From 36
Description: The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: 3 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Score
Arm/Group | Rivaroxaban | Apixaban
Number analyzed (Participants) | 4 | 10
Score | 55.5 [35.6 to 75.4] | 45.6 [25.8 to 80.4]

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events from their baseline visit through their 3-month follow-up visit.
Arm/Group | Rivaroxaban | Apixaban
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 4/8 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=8) | Apixaban (N=11)
Crossover to another anticoagulant (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
PBAC > 100 (Reproductive system and breast disorders) | 2 (5) | 5 (11)
Anticoagulant discontinued for more than 48 hours (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Worsening DVT (Vascular disorders) | 1 (1) | 0 (0)
Bleeding that causes unplanned visit to a healthcare provider (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Terminated secondary to low rate of enrollment despite extraordinary recruitment efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02829957/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02829957/SAP_001.pdf